CLINICAL TRIAL: NCT07307742
Title: Effects of Motor-Focused Exercise Training on Brain Function and Gross Motor Skills in Preschool Children
Brief Title: Motor-Focused Exercise and Brain Development in Preschool Children
Acronym: MoBraD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Normal University (Other)
Responsible Party: Principal Investigator, Liu Bo, Research assistant, Hunan Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HunanNU-2025-532; 2025-532 (Other: Hunan Normal University)
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Child Development; Motor Skills; Neurodevelopment; Brain Function; Executive Function (Cognition)
Keywords: Preschool children; Physical education; Gross motor skills; Motor development; Neurocognitive development; Early childhood education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked to group allocation. Individuals conducting motor skill testing and EEG recordings will not be informed of whether children are in the intervention or control group. Video recordings of motor performance will be independently scored by two raters who are blinded to both group assignment and assessment time point. Data analysts will also remain blinded until the primary analyses are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor-Focused Exercise Training (Experimental): Children will receive structured, motor-focused physical education sessions (30-40 minutes, 3 times per week, for 16 weeks), emphasizing locomotor and object-control skills through playful, game-based activities.
  Interventions: Behavioral: Motor-Focused Physical Education
- Ordinary Physical Education (Active Comparator): Children will continue with their regular kindergarten physical education curriculum (30-40 minutes, 3 times per week, for 16 weeks), focusing on rhythmic movement, free play, and group games.
  Interventions: Behavioral: Ordinary Physical Education

INTERVENTIONS:
Behavioral: Motor-Focused Physical Education — Children will receive structured, motor-focused physical education sessions (30-40 minutes, 3 times per week, for 16 weeks), emphasizing locomotor and object-control skills through playful, game-based activities.
  Arms: Motor-Focused Exercise Training
Behavioral: Ordinary Physical Education — Children will continue with their regular kindergarten physical education curriculum (30-40 minutes, 3 times per week, for 16 weeks), focusing on rhythmic movement, free play, and group games.
  Arms: Ordinary Physical Education

SUMMARY:
This study will test whether a structured motor-focused exercise program can improve both brain function and gross motor skills in preschool children. About 110 children aged 4 to 6 years will be recruited from kindergartens in Changsha, China. Classes will be randomly assigned to receive either (1) motor-focused physical education three times per week for 16 weeks, or (2) ordinary physical education of the same frequency and duration.

The motor-focused program includes playful, game-based activities designed to strengthen locomotor skills (such as running and hopping) and object-control skills (such as throwing and catching). The main outcome will be changes in children's gross motor skills, measured with a standardized motor test (TGMD-3). Brain activity will also be assessed using portable electroencephalography (EEG) during rest and simple tasks related to attention and memory. Parents and teachers will complete short questionnaires about children's behavior and executive function.

The results of this study may provide new insights into how physical education influences both movement skills and brain development in early childhood.

DETAILED DESCRIPTION:
Early childhood is a critical period for both movement and brain development. Learning basic motor skills, such as running, jumping, throwing, and catching, supports later physical activity, health, and learning. At the same time, the brain is rapidly maturing, and experiences that challenge movement and coordination may also strengthen brain systems related to memory, attention, and self-control. However, little is known about how structured physical education influences both motor skill growth and brain function during the preschool years.

This study is designed to test whether a semester-long, motor-focused exercise program can improve gross motor skills and brain activity in preschool children. Approximately 110 children aged 4 to 6 years will be recruited from kindergartens in Changsha, China. Classes will be randomly assigned to one of two groups. The intervention group will participate in structured physical education sessions three times per week, lasting 30-40 minutes, for 16 weeks. These sessions will emphasize locomotor skills (e.g., running, hopping, sliding) and object-control skills (e.g., throwing, catching, kicking), delivered in playful, game-based formats. The control group will continue with ordinary kindergarten physical education, which focuses on rhythmic movement, free play, and group games, also held three times per week.

The primary outcome of the study is gross motor competence, measured using the standardized Test of Gross Motor Development-Third Edition (TGMD-3). Secondary outcomes include brain function assessed with portable electroencephalography (EEG) during rest and during simple tasks measuring attention, memory, and visuomotor control. Parents will complete short questionnaires on executive function in daily life, and teachers will provide ratings of children's behavior and social adjustment. Together, these measures will provide a comprehensive picture of both motor and cognitive development.

The study uses a cluster-randomized controlled trial design, meaning entire kindergarten classes will be randomized as a unit. Outcome assessments will be completed at baseline (before the intervention) and after the 16-week program. Teachers delivering the intervention will receive training and written guidance, and the quality of program delivery will be monitored to ensure fidelity. Motor assessments will be video recorded and scored by independent evaluators who are blinded to group assignment. EEG recordings will follow standardized child-friendly procedures to minimize discomfort.

This trial is among the first to combine structured motor training with direct measures of brain activity in preschool children. By linking improvements in movement skills with changes in brain function, the study aims to provide new insights into how physical education contributes to healthy development in early childhood. Findings may guide schools, teachers, and policymakers in designing more effective physical education programs that promote both physical and cognitive growth.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 6 years enrolled in participating kindergartens in Changsha, China
* Physically healthy and able to safely participate in structured physical education activities
* Written informed consent provided by a parent or legal guardian

Exclusion Criteria:

* Diagnosed neurological, developmental, or musculoskeletal disorders that may interfere with motor performance or EEG measurement
* Currently enrolled in specialized sports or motor-training programs outside of the kindergarten curriculum
* Unable to comply with EEG assessment procedures due to behavioral or sensory intolerance

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Competence (TGMD-3) | Baseline (week 0) and immediately post-intervention (week 16).
  Change in children's gross motor skills measured by the Test of Gross Motor Development-Third Edition (TGMD-3).

SECONDARY OUTCOMES:
EEG Spectral Power | Baseline (week 0) and post-intervention (week 16).
  Change in resting-state EEG spectral power.
Event-Related Potentials (ERP) | Baseline (week 0) and post-intervention (week 16).
  Change in N2 and P3 amplitudes and latencies recorded during Go/No-Go and working memory tasks.
Inhibitory Control | Baseline (week 0) and post-intervention (week 16).
  Accuracy and reaction time on inhibitory control via Go/No-Go.
Working Memory | Baseline (week 0) and post-intervention (week 16).
  Working memory will be assessed according to picture recognition.
Executive Function (Parent Report) | Baseline (week 0) and post-intervention (week 16).
  Parent-rated executive function using the Behavior Rating Inventory of Executive Function-Preschool Version (BRIEF-P).
Behavioral Adjustment (Teacher Report) | Baseline (week 0) and post-intervention (week 16).
  Teacher-rated behavior using the Strengths and Difficulties Questionnaire (SDQ), including domains of prosocial behavior, hyperactivity, and peer relations.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang X, Zhou B. Motor development-focused exercise training enhances gross motor skills more effectively than ordinary physical activity in healthy preschool children: an updated meta-analysis. Front Public Health. 2024 May 21;12:1414152. doi: 10.3389/fpubh.2024.1414152. eCollection 2024. PMID 38835603
- [Result] Lyu W, Thung KH, Huynh KM, Wang L, Lin W, Ahmad S, Yap PT. Functional development of the human cerebellum from birth to age five. Nat Commun. 2025 Jul 10;16(1):6350. doi: 10.1038/s41467-025-61465-y. PMID 40640148
- [Result] Hao Y, Kong L, Wang X, Yu X. The impact of structured motor learning intervention on preschool children's executive functions. Sci Rep. 2025 May 25;15(1):18167. doi: 10.1038/s41598-025-01385-5. PMID 40414940
- [Result] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Result] Chen J, Xiao Y, Xu B, Zhang D. The developmental trajectory of task-related frontal EEG theta/beta ratio in childhood. Dev Cogn Neurosci. 2023 Apr;60:101233. doi: 10.1016/j.dcn.2023.101233. Epub 2023 Mar 16. PMID 36940533
- [Result] Seitz HM, Cottrell BJ, Sturrock RF. A histological study of skin reactions of baboons to Schistosoma mansoni schistosomula. Trans R Soc Trop Med Hyg. 1987;81(3):385-90. doi: 10.1016/0035-9203(87)90144-1. PMID 3120365